CLINICAL TRIAL: NCT03772678
Title: A Phase I Double-blind, Placebo-controlled, Randomized, Single and Multiple Ascending Dose Finding Study to Evaluate the Safety and Pharmacokinetic Profile of LSALT Peptide in Healthy Participants
Brief Title: A Phase I Study to Evaluate LSALT Peptide
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Arch Biopartners Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AB001
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: None - Study is to Determine Safety in Healthy Participants
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacist not blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): 0.9% Saline For SAD and MAD arms.
  Interventions: Other: 0.9% Saline
- Single Ascending Dose - Low Dose (Experimental): LSALT peptide (1mg/mL in 0.9% saline) Single escalating dose - 0.01mg, 0.1mg, 0.3mg, 0.5mg intravenously Escalation to 2.5mg and 5mg doses in next cohorts if no adverse effects are seen after 10-14 days.
  Interventions: Drug: LSALT peptide
- Single Ascending Dose (Experimental): LSALT peptide (1mg/mL in 0.9% saline) Single dose - 1mg intravenously over 2h Escalation to next dose in next participant every 72h if no adverse effects are seen.
  Interventions: Drug: LSALT peptide
- Multiple Ascending Dose (Experimental): LSALT peptide (1mg/mL in 0.9% saline) Dose will be determined based on results of SAD arm. LSALT will be administered intravenously once or twice daily for 3 days.
  Interventions: Drug: LSALT peptide

INTERVENTIONS:
Drug: LSALT peptide — novel 16 amino acid peptide
  Arms: Multiple Ascending Dose; Single Ascending Dose; Single Ascending Dose - Low Dose
Other: 0.9% Saline — saline
  Arms: Placebo

SUMMARY:
A phase I double-blind, placebo-controlled, randomized, single and multiple ascending dose finding study to evaluate the safety and pharmacokinetic profile of LSALT peptide in healthy participants

ELIGIBILITY:
Inclusion Criteria:

* No prior history of major organ or systemic disease including diabetes, hypertension, kidney, heart or liver disease. Participants with childhood asthma are acceptable.
* Normal hematology, clinical chemistry and urinalysis parameters at screening, unless not deemed clinically significant by the investigator.
* Body Mass Index (BMI) between 18 kg/m2 and 32 kg/m2 (inclusive)
* Taking no prescription medications 2 weeks prior to admission or over-the-counter medications 7 days prior to admission. Occasional use of paracetamol or ibuprofen (up to 1000 mg and 400 mg/day respectively) are acceptable. Routine vitamins and supplements are permissible at the discretion of the investigator.
* Able to allow intravenous medication to be administered.
* Males (along with their female partners) and females of childbearing potential (defined as a female who is not menopausal or surgically sterilized) must be willing to use an acceptable method of birth control during heterosexual activities including a condom and a second highly effective method (i.e., hormonal contraceptive, intra-uterine device) or abstinence for the duration of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Males should continue with the aforementioned contraception for 90 days after the last dose and females should continue with the aforementioned contraception for 60 days after last dose.
* Able to understand and willing to sign an ethics committee-approved written informed consent document
* Non-smokers. Social and light smokers of up to 10 cigarettes per day who can abstain from smoking during the confinement period and have no evidence of underlying lung disease (bronchitis, COPD or reactive airways disease).
* Willing to remain abstinent from alcohol 24 hours prior to admission and until after the confinement period in the unit.

Exclusion Criteria:

* A history of cardiovascular disease, diabetes or hypertension (>150/90 after 5 minutes sitting), significant neurological, pulmonary (including asthma), hepatic, rheumatic, autoimmune, haematological, metabolic or renal disorder.
* Prescription medications are prohibited. No prescription medications 2 weeks prior to admission or over-the-counter medications 7 days prior to admission. Occasional use of paracetamol or ibuprofen (up to 1000 mg and 400 mg/day respectively) are acceptable. Routine vitamins and supplements are permissible at the discretion of the investigator.
* Any moderate or severe allergies, including anaphylaxis, to food, drugs or environmental allergens. Mild allergies such as hayfever may be included.
* Females who are pregnant or lactating. Women of childbearing potential must have a negative pregnancy test within 14 days of study initiation and at baseline.
* Consumption of caffeine 48 hours prior to start of study treatment and whilst confined to the unit.
* History of any psychiatric illness or psychological disorder which may impair the ability to provide written informed consent or participate in the study
* Clinically significant abnormal laboratory value at screening as determined by the Investigator.
* Participant is sero-positive to HIV-1 or HIV-2, HCV or HBV.
* History or presence of alcoholism within two years prior to the first study drug administration or drugs of abuse unless it can be explained to the satisfaction of the investigator that it is due to a standard dose of a prescribed medication and that an adequate wash-out will occur prior to admission.
* No findings on clinical examination that, in the opinion of the investigator, could compromise the safety of the participant or the results of the study.
* Blood donation or significant blood loss within 60 days prior to the first study drug administration.
* Administration of investigational product in another trial within 30 days prior to the first study drug administration or five half-lives, whichever is longer.
* Surgery within the past 3 months prior to the first study drug administration determined by the PI to be clinically relevant.
* Active malignancy or history of malignancy in the past 5 years.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Ltd., Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LSALT Peptide - 0.01mg: LSALT peptide (1mg/mL in 0.9% saline) single dose intravenously.
  Escalation to 0.1mg dose in next cohort if no adverse effects are seen after 3 days.
  LSALT peptide: novel 16 amino acid peptide
- LSALT Peptide - 0.1mg: LSALT peptide (1mg/mL in 0.9% saline) single dose intravenously.
  Escalation to 0.3mg dose in next cohort if no adverse effects are seen after 3 days.
  LSALT peptide: novel 16 amino acid peptide
- LSALT Peptide - 0.3mg: LSALT peptide (1mg/mL in 0.9% saline) single dose intravenously.
  Escalation to 0.5mg dose in next cohort if no adverse effects are seen after 3 days.
  LSALT peptide: novel 16 amino acid peptide
- LSALT Peptide - 0.5mg: LSALT peptide (1mg/mL in 0.9% saline) single dose intravenously.
  Escalation to 1.0mg dose in next cohort if no adverse effects are seen after 10-14 days.
  LSALT peptide: novel 16 amino acid peptide
- LSALT Peptide - 1.0mg: LSALT peptide (1mg/mL in 0.9% saline) single dose - 1.0mg intravenously over 2h.
  Escalation to next dose (2.5mg) in next cohort if no adverse effects are seen.
  LSALT peptide: novel 16 amino acid peptide
- LSALT Peptide - 2.5mg: LSALT peptide (1mg/mL in 0.9% saline) single dose - 2.5mg intravenously over 2h.
  Escalation to next dose (5.0mg) in next cohort if no adverse effects are seen.
  LSALT peptide: novel 16 amino acid peptide
- LSALT Peptide - 5.0mg: LSALT peptide (1mg/mL in 0.9% saline) single dose - 5.0mg intravenously over 2h.
  Escalation to multiple ascending dose cohort if no adverse effects are seen.
  LSALT peptide: novel 16 amino acid peptide
- Placebo - Single Dose: 0.9% saline as placebo for single dose cohorts (1.0mg, 2.5mg, 5.0mg)
- LSALT Peptide - 1.0mg, Multiple Ascending Dose: LSALT peptide (1mg/mL in 0.9% saline) single dose (1.0mg) per day intravenously over 2h.
  LSALT will be administered intravenously once daily for 3 days.
  LSALT peptide: novel 16 amino acid peptide
- LSALT Peptide - 2.5mg, Multiple Ascending Dose: LSALT peptide (1mg/mL in 0.9% saline) single dose (2.5mg) per day intravenously over 2h.
  LSALT will be administered intravenously once daily for 3 days.
  LSALT peptide: novel 16 amino acid peptide
- LSALT Peptide - 5.0mg, Multiple Ascending Dose: LSALT peptide (1mg/mL in 0.9% saline) single dose (5.0mg) per day intravenously over 2h.
  LSALT will be administered intravenously once daily for 3 days.
  LSALT peptide: novel 16 amino acid peptide
- Placebo - Multiple Ascending Dose: 0.9% saline as placebo for multiple ascending dose cohorts (1.0mg, 2.5mg, 5.0mg)
Period: Overall Study
Arm/Group | LSALT Peptide - 0.01mg | LSALT Peptide - 0.1mg | LSALT Peptide - 0.3mg | LSALT Peptide - 0.5mg | LSALT Peptide - 1.0mg | LSALT Peptide - 2.5mg | LSALT Peptide - 5.0mg | Placebo - Single Dose | LSALT Peptide - 1.0mg, Multiple Ascending Dose | LSALT Peptide - 2.5mg, Multiple Ascending Dose | LSALT Peptide - 5.0mg, Multiple Ascending Dose | Placebo - Multiple Ascending Dose
Started | 1 | 1 | 1 | 1 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 1 | 1 | 1 | 1 | 5 | 5 | 6 | 5 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo - Multiple Ascending Dose: 0.9% saline as placebo for multiple ascending dose cohorts
- Total: Total of all reporting groups
Arm/Group | LSALT Peptide - 0.01mg | LSALT Peptide - 0.1mg | LSALT Peptide - 0.3mg | LSALT Peptide - 0.5mg | LSALT Peptide - 1.0mg | LSALT Peptide - 2.5mg | LSALT Peptide - 5.0mg | Placebo - Single Dose | LSALT Peptide - 1.0mg, Multiple Ascending Dose | LSALT Peptide - 2.5mg, Multiple Ascending Dose | LSALT Peptide - 5.0mg, Multiple Ascending Dose | Placebo - Multiple Ascending Dose | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 1 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 52
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 1 | 3 | 2 | 3 | 1 | 2 | 3 | 2 | 21
  Male | 0 | 0 | 0 | 0 | 5 | 3 | 4 | 3 | 5 | 4 | 3 | 4 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 3 | 3 | 1 | 2 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 0 | 1 | 1 | 1 | 4 | 3 | 4 | 5 | 3 | 3 | 4 | 4 | 33
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety Evaluation
Description: To determine the safety and tolerability of 3 single and multiple ascending doses of LSALT peptide (1.0mg, 2.5mg, 5.0mg) in healthy participants.
Time Frame: Within 21 days
Population: The Safety Population was comprised of all randomised subjects who received any amount of study drug in the single ascending dose and multiple ascending dose cohorts and were based on the actual treatment received, if this differs from that to which the subject was randomised. The Safety Population was used for the summaries of all safety tolerability.
Measure: Number; unit: participants
Arm/Group | LSALT Peptide - 0.01mg | LSALT Peptide - 0.1mg | LSALT Peptide - 0.3mg | LSALT Peptide - 0.5mg | LSALT Peptide - 1.0mg | LSALT Peptide - 2.5mg | LSALT Peptide - 5.0mg | Placebo - Single Dose | LSALT Peptide - 1.0mg, Multiple Ascending Dose | LSALT Peptide - 2.5mg, Multiple Ascending Dose | LSALT Peptide - 5.0mg, Multiple Ascending Dose | Placebo - Multiple Ascending Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  At least One TEAE |  |  |  |  | 3 | 1 | 6 | 2 | 5 | 4 | 2 | 5
  At least One Severe or Life-threatening TEAE |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  At least One Study Drug-related TEAE |  |  |  |  | 0 | 0 | 2 | 1 | 3 | 1 | 1 | 1
  At least One Serious TEAE |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  At least One Serious Study Drug-related TEAE |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Discontinuation due to TEAE |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Death |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetic Evaluation
Description: To evaluate the PK and pharmacodynamics (PD) of LSALT peptide in healthy participants.
Time Frame: Within 21 days
Population: The PK Concentration Population was comprised of all subjects who received any amount of LSALT, who had at least 1 quantifiable PK concentration and was based on the actual treatment received, if this differs from that to which the subject was randomized. Subjects who received only placebo was excluded from the PK Concentration Population. The PK Concentration Population was used for the summaries of all PK concentration data.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- LSALT Peptide - 5.0mg: LSALT peptide (1mg/mL in 0.9% saline) single dose - 5.0mg intravenously over 2h.
  LSALT peptide: novel 16 amino acid peptide
Arm/Group | LSALT Peptide - 5.0mg | LSALT Peptide - 5.0mg, Multiple Ascending Dose
Number analyzed (Participants) | 6 | 6
hours
  T1/2 (h) | 0.41 (0.147) | 0.21 (0.075)
  Tmax (h) | 1.33 (0.6) | 1.17 (0.516)

ADVERSE EVENTS:
Time Frame: For Low Dose cohort - study subjects were monitored for 3 days For SAD cohort - study subjects were monitored for 7 days For MAD cohort - study subjects were monitored for 21 days
Arm/Group | LSALT Peptide - 0.01mg | LSALT Peptide - 0.1mg | LSALT Peptide - 0.3mg | LSALT Peptide - 0.5mg | LSALT Peptide - 1.0mg | LSALT Peptide - 2.5mg | LSALT Peptide - 5.0mg | Placebo - Single Dose | LSALT Peptide - 1.0mg, Multiple Ascending Dose | LSALT Peptide - 2.5mg, Multiple Ascending Dose | LSALT Peptide - 5.0mg, Multiple Ascending Dose | Placebo - Multiple Ascending Dose
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 3/6 | 1/6 | 6/6 | 2/6 | 5/6 | 4/6 | 2/6 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LSALT Peptide - 0.01mg (N=1) | LSALT Peptide - 0.1mg (N=1) | LSALT Peptide - 0.3mg (N=1) | LSALT Peptide - 0.5mg (N=1) | LSALT Peptide - 1.0mg (N=6) | LSALT Peptide - 2.5mg (N=6) | LSALT Peptide - 5.0mg (N=6) | Placebo - Single Dose (N=6) | LSALT Peptide - 1.0mg, Multiple Ascending Dose (N=6) | LSALT Peptide - 2.5mg, Multiple Ascending Dose (N=6) | LSALT Peptide - 5.0mg, Multiple Ascending Dose (N=6) | Placebo - Multiple Ascending Dose (N=6)
General Disorders and Administration Site Conditions (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 1 | 6 | 2 | 3 | 3 | 0 | 0
Infections and Infestations (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Nervous System Disorders (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 3 | 0 | 0
Gastrointestinal Disorders (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Respiratory, Thoracic, and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular Disorders (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye Disorders (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (3):
  • Study Protocol (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT03772678/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT03772678/SAP_001.pdf
  • Informed Consent Form (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT03772678/ICF_002.pdf